CLINICAL TRIAL: NCT05698888
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of VP301 in Patients With Relapsed or Refractory Multiple Myeloma, Lymphoma, or Solid Tumors
Brief Title: Study of VP301 in Patients With Multiple Myeloma, Lymphoma, or Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Virtuoso BINco, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VP301-001
Record Dates: First submitted 2022-12-12; First posted 2023-01-26 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumors, Adult; Multiple Myeloma; Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma

STUDY DESIGN:
Intervention Model Description: Following completion of the dose escalation phase of the study and determination of maximum tolerated dose or recommended phase 2 dose, patients will be enrolled into dose expansion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VP301 (Dose Escalation) (Experimental): Eligible patients will receive VP301 administered as an IV infusion weekly for 6 weeks then every 2 weeks. Patients will be enrolled into escalating dose levels during the Dose Escalation period of the study.
  Interventions: Drug: VP301
- VP301 (Dose Expansion) (Experimental): Eligible patients will receive VP301 administered as an IV infusion weekly for 6 weeks then every 2 weeks. Patients will receive the maximum tolerated dose or recommended phase 2 dose during the Dose Expansion period of the study.
  Interventions: Drug: VP301

INTERVENTIONS:
Drug: VP301 — VP301 is an afucosylated humanized Fc-modified immunoglobulin G1 (IgG1) bispecific antibody targeting CD38 and ICAM-1.

SUMMARY:
This study will test the safety, tolerability, and pharmacokinetics of VP301 in patients with relapsed or refractory multiple myeloma, lymphoma, or solid tumors.

DETAILED DESCRIPTION:
This study will test the safety, tolerability, and pharmacokinetics of VP301 in patients with relapsed or refractory multiple myeloma, lymphoma, or solid tumors. This study will be conducted in two parts:

Dose Escalation - This part will evaluate increasing doses of VP301 to identify the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D). The first patient enrolled on the study will receive the lowest dose of VP301. Once this dose is shown to be safe, an additional patient will be enrolled at the next higher dose. Patients will continue to be enrolled into either single or multiple patient groups receiving increasing doses until the MTD or RP2D is reached.

Dose Expansion - Patients with relapsed myeloma and lymphoma will be enrolled and treated with VP301 at the MTD or RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of a refractory solid tumor, refractory myeloma or lymphoma with measurable or evaluable disease
* Patients must have progressed following all therapies of known, potential clinical benefit, or for whom treatments of known clinical benefit are contraindicated.
* Adequate kidney, liver, and hematologic function
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2

Exclusion Criteria:

* Active brain metastases and history of leptomeningeal metastases.
* Myeloma patients with plasmacytoma as only measurable disease
* Non-secretory myeloma
* Patients with advanced metastatic, symptomatic, visceral spread who are at risk of life-threatening complications
* Active or chronic, uncontrolled bacterial, viral, or fungal infection(s)
* Abnormal ECG
* Has clinically significant cardiovascular disease
* Additional active malignancy that may confound the assessment of the study endpoints
* Pregnancy or lactation
* Known seropositivity for HIV (human immunodeficiency virus) or active hepatitis B or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Occurrence of General Toxicity | through study completion, an average of 30 months
  Incidence of treatment-emergent serious AEs including toxicity and change from baseline in safety parameters
Occurrence of Dose Limiting Toxicity | Over the first 21 days of VP301 dosing
  Incidence of dose limiting toxicity during cycle 1 of dose escalation

SECONDARY OUTCOMES:
Serum concentrations of VP301 | through study completion, an average of 30 months
  Change from baseline in serum levels
Antidrug and neutralizing antibodies | through study completion, an average of 30 months
  Change from baseline in serum levels
Objective response | through study completion, an average of 30 months
  Assessed by IMWG for multiple myeloma, the Lugano criteria for lymphoma or RECIST 1.1 for solid tumors
Best response | through study completion, an average of 30 months
  Assessed by IMWG for multiple myeloma, the Lugano criteria for lymphoma or RECIST 1.1 for solid tumors
Time to response and duration of response | through study completion, an average of 30 months
  Assessed by IMWG for multiple myeloma or the Lugano criteria for lymphoma
Progression-free survival | through study completion, an average of 30 months
  Assessed by IMWG for multiple myeloma or the Lugano criteria for lymphoma

OTHER OUTCOMES:
Tumor expression | through study completion, an average of 30 months
  Evaluate ICAM-1 and CD38 expression with clinical outcomes
Immunoglobulins | through study completion, an average of 30 months
  Evaluate quantitative immunoglobulins with clinical outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- NEXT Oncology, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No